CLINICAL TRIAL: NCT00617773
Title: A PHASE II TRIAL OF Hu3S193 THERAPY FOR PATIENTS WITH PLATINUM REFRACTORY OR PLATINUM RESISTANT EPITHELIAL OVARIAN, PRIMARY PERITONEAL AND FALLOPIAN TUBE CANCER
Brief Title: Hu3S193 in Treating Women With Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recepta Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCPOv01-06; RCP-Ov-01.06 (Other: Recepta Biopharma)
Record Dates: First submitted 2008-02-15; First posted 2008-02-18 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hu3S193 (Experimental)
  Interventions: Biological: hu3S193

INTERVENTIONS:
Biological: hu3S193 — 20 mg/m2, intravenous, weekly for a maximum of 3 cycles (of 8 weeks each)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as Hu3S193, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well Hu3S193 works in treating patients with ovarian epithelial cancer, fallopian tube cancer, or peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of monoclonal antibody Hu3S193 in women with platinum-resistant/refractory ovarian, fallopian tube, or primary peritoneal cancer, based on RECIST criteria (Response Evaluation Criteria in Solid Tumors).

Secondary

* To determine the safety of the study drug.
* To determine the drug pharmacokinetics when administered in multiple weekly injections.

Exploratory analysis

* Clinical Benefit (objective response rate + tumor stabilization).
* Progression Free Survival (PFS).
* Duration of Response.
* Overall Survival.
* 12-month survival rate.

OUTLINE: This is a multicenter study.

Patients receive monoclonal antibody Hu3S193 IV over 1 hour once weekly in weeks 1-8. Treatment repeats every 8 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed monthly.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Progressive disease
  * Disease must express Lewis-Y antigen documented by immunohistochemistry in archived or fresh primary or metastatic tumor biopsies
* Measurable disease, including at least one measurable lesion, according to RECIST criteria or CA-125 (Cancer Antigen-125) > 2 times upper normal limit

  * Pleural effusion, ascites, bone metastases, and lesions located in previously irradiated areas are not considered measurable
* Disease must be considered platinum-refractory or resistant, meeting any of the following criteria:

  * Platinum-refractory defined as progression during the initial platinum-based chemotherapy regimen or failure to achieve a complete response (e.g., stable disease or partial response) with evidence of progressive disease (by physical examination, radiological exams, or CA-125) during the initial platinum-based chemotherapy
  * Platinum-resistant defined as recurrence within six months of completion of the initial platinum-based regimen (primary platinum-resistance) or recurrence after six months of completion of the initial platinum-based regimen (still considered platinum-sensitive, but incurable by any approach, that will progress to a secondary platinum-resistance scenario) and failure to ≥ 1 re-induction with a platinum-based regimen (secondary platinum-resistance)
* No high tumor burden, as assessed by the investigator
* No rapidly progressing disease, as assessed by clinical evaluation
* No known CNS (Central Nervous System) involvement by tumor

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status > 70%
* Life expectancy ≥ 12 weeks
* ANC (absolute neutrophil count) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum bilirubin ≤ 2.0 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN if with liver metastases)
* Creatinine ≤ 2.0 mg/dL
* Prothrombin time < 1.3 times control
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* NYHA (New York Heart Association) class III or IV heart disease
* Clinically significant arrhythmias by ECG
* Myocardial infarction within the past 6 months
* Any other serious illness, including any of the following:

  * Severe ascites
  * Severe active infections requiring antibiotics
  * Bleeding disorders
  * Chronic inflammatory bowel disease
  * Diseases that might interfere with the collection of accurate results from this study
* Positive for human anti-human antibodies
* Prior history of tumor (excluding adequately treated nonmelanoma skin cancer or carcinoma in situ of the uterine cervix)
* Uncontrolled hypercalcemia (i.e., > 11.5 mg/dL)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the toxic effects of any prior therapy
* No concurrent systemic steroids or immunosuppressant agents
* No more than 1 prior non-platinum-containing regimen for the treatment of platinum-resistant/refractory disease

  * Patients who receive 2 or more different non-platinum-containing chemotherapy regimens for platinum-resistant/refractory disease are not eligible
* More than 4 weeks since prior and no other concurrent chemotherapy, radiotherapy, radiopharmaceuticals (e.g., ^32P), biological therapy, anti-estrogen therapy (including tamoxifen), immunotherapy, or surgery
* More than12 weeks since prior investigational agent
* No prior treatment with a murine or humanized antibody and/or antibody fragment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oren Smaletz, MD, Study Chair — Recepta Biopharma
Locations (8):
- Brazil (8):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Hospital da Baleia, Minas Gerais
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital das Clinicas FMUSP, São Paulo
  - Hospital Sirio-Libanes, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo

REFERENCES:
- [Derived] Smaletz O, Diz MD, do Carmo CC, Sabbaga J, Cunha-Junior GF, Azevedo SJ, Maluf FC, Barrios CH, Costa RL, Fontana AG, Madrigal V, Wainstein AJ, Yeda FP, Alves VA, Moro AM, Blasbalg R, Scott AM, Hoffman EW. A phase II trial with anti-Lewis-Y monoclonal antibody (hu3S193) for the treatment of platinum resistant/refractory ovarian, fallopian tube and primary peritoneal carcinoma. Gynecol Oncol. 2015 Aug;138(2):272-7. doi: 10.1016/j.ygyno.2015.05.023. Epub 2015 May 27. PMID 26026738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a brazilian, multicentric clinical trial. From June 20, 2008 to July 13, 2010 (recruitment period of 24 months) a total of 51 patients were screened for this study, of whom 31 were considered eligible and received at least one dose of the investigational product and 20 were considered non-eligible.
Pre-assignment Details: Patients were considered included in the study on the day of the first investigational product administration after investigator assured that patients met all the inclusion criterions and none of the exclusion criterions.
Groups:
- hu3S193: hu3S193 : 20 mg/m2, intravenous, weekly for a maximum of 3 cycles (of 8 weeks each)
Period: Overall Study
Arm/Group | hu3S193
Started | 31
Completed | 7 (Patients COMPLETED were evaluated as having no disease progression at the end of cycle 3.)
Not Completed | 24
Not completed — Physician Decision | 1
Not completed — Lack of compliance with the protocol | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Progressive disease | 19
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The baseline descriptive analyses were performed for the safety population. Lewis Y antigen expression and blood type were also analyzed for this population.
Arm/Group | hu3S193
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 31
Expression of the Lewis Y antigen in tumor tissue [Number; unit: participants] — Expression of Lewis Y was investigated by immunohistochemistry on primary or metastatic tumor biopsies. To determine Lewis Y expression levels, a semi-quantitative approach was used, which considered cytoplasm and membrane compartments independently. The score taken into account was from the higher expression observed, either cytoplasm or membrane.
  Participants with positive expression of Lewis Y in tumor were scored, according to the percentage of positively stained cells, into the following categories: +4 (>75% positive cells); +3 (51 to 75%); +2 (26 to 50%); and +1 (1 to 25%).
  participants
    Positive (+1) | 14
    Positive (+2) | 6
    Positive (+3) | 8
    Positive (+4) | 3
ABO blood type [Number; unit: participants]
  Type A | 11
  Type B | 1
  Type AB | 2
  Type O | 17

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Best response recorded from the start of treatment until disease progression/recurrence. Includes all patients evaluable for efficacy, regardless of used criteria: RECIST or CA-125 (Cancer Antigen 125).
  Evaluation of target lesions: Complete Response (CR), resolution of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD sum) of target lesions, taking as reference the baseline LD sum; Progressive Disease (PD), a 20% increase in LD sum of target lesions or the appearance of new lesion(s); Stable Disease (SD), no sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD. Evaluation of non-target lesions: CR, resolution of all non-target lesions and normalization of CA-125 level; SD, persistence of one or more non-target lesions and/or maintenance of CA-125 level above the normal limits; PD, appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: From start of study treatment until the end of Cycle 1 (8 weeks), Cycle 2 (16 weeks) or Cycle 3 (24 weeks).
Population: All patients enrolled in the study that received at least 4 doses of investigational product were considered to the efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | hu3S193
Number analyzed (Participants) | 26
participants
  Complete response | 0
  Partial response | 0
  Stable disease | 13
  Disease progression | 11
  Unknown | 2

2. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: A listing of all adverse events is located in the Reported Adverse Event module.
Time Frame: From the first dose of investigational product up to 30 days after the last dose of investigational product
Population: All patients enrolled in the study that received at least 1 dose of investigational product were considered for safety evaluation.
Measure: Number; unit: participants
Arm/Group | hu3S193
Number analyzed (Participants) | 31
participants
  Adverse Events | 31
  Serious Adverse Events | 9

3. Secondary Outcome: Number of Participants With Adverse Events Reasonably Related to the Investigational Product (Incidence Greater Than 5%).
Description: Adverse events with possible, probable or definite relationship to the investigational product were considered to be reasonably related.
Time Frame: From the first dose of investigational product up to 30 days after the last dose of investigational product
Measure: Number; unit: participants
Arm/Group | hu3S193
Number analyzed (Participants) | 31
participants
  Adverse event: Nausea | 5
  Adverse event: Fatigue | 4
  Adverse event: Diarrhoea | 3
  Adverse event: Hypersensitivity | 3
  Adverse event: Hypertension | 3
  Adverse event: Pyrexia | 3
  Adverse event: Constipation | 2
  Adverse event: Dry mouth | 2
  Adverse event: Haemoglobin abnormal | 2
  Adverse event: Tremor | 2
  Adverse event: Urticaria | 2

4. Secondary Outcome: Mean Cmax and Cmin of Hu3S193 Relating to the First 4 Doses.
Description: Cmax = Peak (post-dosing) IP (Investigational Product) plasma concentration. Cmin = Trough (pre-dosing) IP plasma concentration (Cmin). Plasma concentration of Hu3S193 expressed in µg/mL.
Time Frame: Pre-dose (within 10 minutes) and Post-dose (5 minutes after completion of infusion) on weeks 1, 2, 3, and 4 of Cycle 1.
Population: All patients enrolled in the study that received at least 4 doses of investigational product were considered to this analysis.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | hu3S193
Number analyzed (Participants) | 26
µg/mL
  Mean Cmax of Hu3S193 | 16.7 (3.7)
  Mean Cmin of Hu3S193 | 2.1 (1)

5. Secondary Outcome: Mean Cmax and Cmin of Hu3S193 Relating to the First 8 Doses
Description: Cmax = Peak (post-dosing) IP plasma concentration. Cmin = Trough (pre-dosing) IP plasma concentration (Cmin). Plasma concentration of Hu3S193 expressed in µg/mL.
Time Frame: Pre-dose (within 10 minutes) and Post-dose (5 minutes after completion of infusion) on weeks 1, 2, 3, 4, 5, 6, 7 and 8 of Cycle 1.
Population: All patients enrolled in the study that received at least 8 doses of investigational product were considered to this analysis.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | hu3S193
Number analyzed (Participants) | 17
µg/mL
  Mean Cmax of Hu3S193 | 10.9 (4.7)
  Mean Cmin of Hu3S193 | 2.3 (0.8)

6. Other Pre Specified Outcome: Clinical Benefit
Description: The clinical benefit was calculated considering all patients with objective response rate (CR + PR) or stable disease (SD) for at least 24 weeks according RECIST or CA-125 if patients were non-assessable or when assessment by RECIST was unknown.
  Clinical benefit = 100% x (Number of patients with objective response + Number of patients with stable disease for at least 24 weeks) / Number of patients included in the efficacy population.
  The evaluation of target and non-target lesions is described at the Outcome Measure titled "Best Overall Response". CR: Complete Response; PR: Partial Response; SD: Stable Disease.
Time Frame: From start of study treatment until the end of Cycle 3 (24 weeks).
Population: All patients enrolled in the study that received at least 4 doses of investigational product and that were evaluable for response were considered to this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | hu3S193
Number analyzed (Participants) | 24
percentage of participants | 25.0 [9.77 to 46.71]

7. Other Pre Specified Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the duration of time from start of treatment to time of disease progression.
Time Frame: From the first day of the investigational product administration until documentation of disease progression or death due to any cause (whichever occurred first). An average of 16.5549 weeks.
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | hu3S193
Number analyzed (Participants) | 26
weeks | 8.4286 [4.1429 to 87.0000]

8. Other Pre Specified Outcome: Overall Survival
Description: Measured from the beginning of therapy until the date of death or for patients without a known date of death, they will be censored at the date they were last known to be alive.
Time Frame: From start of study treatment until death or the date that patients were last known to be alive. An average of 56.126 weeks.
Population: as for outcome 4
Measure: Median (Full Range); unit: weeks
Arm/Group | hu3S193
Number analyzed (Participants) | 26
weeks | 67.214 [4.714 to 131.143]

9. Other Pre Specified Outcome: 12-Month Survival Rate
Description: Rate of patients alive 12 months after starting therapy with the investigational product.
Time Frame: 12 months from the start of study treatment.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | hu3S193
Number analyzed (Participants) | 26
percentage of participants | 57.7 [38.7 to 76.7]

10. Post Hoc Outcome: Progression Free Survival in Patients With and Without Ascites at Baseline
Description: as for outcome 7
Time Frame: From the first day of the investigational product administration until documentation of disease progression or death due to any cause (whichever occurred first) while the patient was on treatment, non-treatment period, or during the long-term follow-up.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | hu3S193
Number analyzed (Participants) | 26
weeks
  PFS in patients with ascites at baseline (n=9) | 6.0000 [4.7143 to 8.2857]
  PFS in patients without ascites at baseline (n=17) | 16.1429 [7.1429 to 32.0000]

11. Post Hoc Outcome: Progression Free Survival in Patients With and Without Visceral Disease at Baseline
Description: as for outcome 7
Time Frame: as for outcome 10
Population: All patients enrolled in the study that received at least 4 doses of investigational product and that were assessed for visceral disease at baseline were considered for this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | hu3S193
Number analyzed (Participants) | 25
weeks
  PFS in patients with visceral disease (n=5) | 6.1429 [4.1429 to 28.0000]
  PFS in patients without visceral disease (n=20) | 8.9286 [5.4286 to 18.2857]

12. Post Hoc Outcome: Progression Free Survival in Patients Without Ascites and no Visceral Disease at Baseline Versus Patients With Ascites and/or Visceral Disease at Baseline
Description: as for outcome 7
Time Frame: as for outcome 10
Population: All patients enrolled in the study that received at least 4 doses of investigational product and that were assessed for visceral disease and ascites at baseline were considered for this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | hu3S193
Number analyzed (Participants) | 25
weeks
  Without ascites and no visceral disease (n=13) | 16.1429 [7.1429 to 32.0000]
  With ascites and/or visceral disease (n=12) | 6.0714 [4.7143 to 8.2857]

ADVERSE EVENTS:
Time Frame: From the first dose of investigational product up to 30 days after the last dose of investigational product.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings.
Arm/Group | hu3S193
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hu3S193 (N=31)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Asthenia; Performance status decreased (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hu3S193 (N=31)
Nausea (Gastrointestinal disorders) | 13 (21)
Vomiting (Gastrointestinal disorders) | 13 (26)
Abdominal pain (Gastrointestinal disorders) | 12 (16)
Constipation (Gastrointestinal disorders) | 10 (14)
Diarrhoea (Gastrointestinal disorders) | 10 (14)
Fatigue (General disorders) | 8 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pyrexia (General disorders) | 6 (8)
Anorexia (Gastrointestinal disorders) | 5 (10)
Haemoglobin abnormal (Investigations) | 5 (9)
Influenza like illness (General disorders) | 5 (6)
Tremor (Nervous system disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Headache (Nervous system disorders) | 4 (5)
Oedema peripheral (General disorders) | 4 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (6)
Chest pain (General disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Hypersensitivity (Immune system disorders) | 3 (5)
Hypertension (Vascular disorders) | 3 (10)
Insomnia (Psychiatric disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Catheter site pain (General disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less